CLINICAL TRIAL: NCT00348075
Title: A Singapore Study To Evaluate The Efficacy OF Neurovision'S NVC™- Vision Correction Technology For The Visual Improvement In Subjects With Low Or Moderate Adult Myopia
Brief Title: A Singapore Study to Assess How Neurovision Improve the Vision of Adults With Low to Moderate Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Defence Medical Research Institute, Singapore Armed Forces (Unknown); NeuroVision (Industry)
Responsible Party: Donald Tan, Singapore Eye Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R330/23/2003
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Myopia
Keywords: Neurovision; Adult myopia; Therapy
MeSH Terms: conditions — Myopia

ARMS (1):
- Neurovision (Experimental)
  Interventions: Device: Neurovision

INTERVENTIONS:
Device: Neurovision

SUMMARY:
To evaluate the efficacy of NeuroVision NVC vision correction technology to improve the vision of subjects with Low and Moderate Myopia in Asian eyes in Singapore

DETAILED DESCRIPTION:
NeuroVision has developed a novel vision correction technology, which is a scientifically based treatment to improve vision based on new principles of visual psychophysics. NeuroVision NVC Vision Correction Technology is a non-invasive, patient-specific treatment based on visual stimulation and facilitation of neural connections responsible for vision. The treatment involves a programmed series of interactive visual exercises in front of a computer, and does not involve any form of prescription medications, or surgical treatment.

The technology has been proven in both Israel and Singapore's pilot study to work for myopia -1.50D and below.

This study is a clinical trial for Singapore Ministry of Defence personnel to evaluate the efficacy of this treatment beyond the proven myopia range. There will be 2 phases in the study; Phase 1 will include low myopes from -0.50D to -1.50D while Phase 2 covers moderate myopes from -1.75D to -3.00D. Subjects will be randomised into treatment and placebo group in the ratio of 3:1.

A randomized double masked controlled trial conducted in 2 Phases:

Phase I will involve 140 study subjects with low myopia randomized in a 3:1 randomization to receive NVC treatment versus placebo treatment.

It is assumed that the withdrawal rate will not exceed 20%, so that at least 112 study subjects will complete the treatment phase.

Interim analysis with stopping rule will be conducted after 3/4 of the patients complete the treatment phase.

Phase II will involve 180 study subjects with moderate myopia randomized in a 3:1 randomization to receive NVC treatment versus placebo treatment.

The 2 phases will be separate RCTs, with recruitment of Phase II subjects subsequent to completion of Phase I NVC treatments.

ELIGIBILITY:
Inclusion Criteria for Phase I NVC-AM1 (Low Myopia):

1. The subject's cycloplegic spherical equivalence in the worst eye is within the range of -0.50DS to -1.50DS of myopia, and astigmatism does not exceed 0.75DC in either eye.
2. The subject's refractive status is stable, with no increase beyond 0.5D in sphere or cylinder over the last six months.
3. The subject's age is between 17-55 years.
4. The subject's uncorrected visual acuity in both eyes should be between 0.1 and 0.7 logMAR.
5. The subject's best corrected visual acuity 0.05 LogMar (either eye)
6. The subject is cognitively intact and is able to follow multiple step instructions.
7. The subject is able to cease contact lens wear from Baseline examination onwards until the end of the treatment period. The subject is able to cease contact lens wear for at least a week before attending the Baseline examination, Post-treatment evaluation and Persistence evaluation.
8. The subject is able and willing to attend all study sessions and visits at the required frequency:

   1. The total number of treatments is individual, approximately 30.
   2. The required pace for the treatment sessions is at least 3 sessions per week.
   3. No foreseen interruptions longer than 2 weeks during the treatment course.
9. Subject (or subject's parent/legal guardian if subject is less than 21 years of age at study entry) agrees to sign the Informed Consent Form (See Appendix D)
10. Manifest spherical equivalence - not more than 1.0Ds difference from cycloplegic spherical equivalence
11. Unaided VA difference between both eyes is less than 0.3 logMAR
12. The patient is very keen to improve unaided vision and to decrease the dependency on eye glasses

Inclusion criteria for Phase II NVC-AM2 (Moderate Myopia):

1. The subject's cycloplegic spherical equivalence in the worst eye is within the range of -1.750DS to -3.0DS of myopia, and astigmatism does not exceed 0.75DC in either eye.
2. The subject's refractive status is stable, with no increase beyond 0.5D in sphere or cylinder over the last six months.
3. The subject's age is between 17-55 years.
4. The subject's uncorrected visual acuity in the worst eye should not exceed 1.0 logMAR.
5. The subject's best corrected visual acuity 0.05 LogMar (either eye)
6. The subject is cognitively intact and is able to follow multiple step instructions.
7. The subject is able to cease contact lens wear from Baseline examination onwards until the end of the treatment period. The subject is able to cease contact lens wear for at least a week before attending the Baseline examination, Post-treatment evaluation and Persistence evaluation.
8. The subject is able and willing to attend all study sessions and visits at the required frequency:

   1. The total number of treatments is individual, approximately 30.
   2. The required pace for the treatment sessions is at least 3 sessions per week.
   3. No foreseen interruptions longer than 2 weeks during the treatment course.
9. Subject (or subject's parent/legal guardian if subject is less than 21 years of age at study entry) agrees to sign the Informed Consent Form (See Appendix D)

Exclusion Criteria (for both Phase I and II):

1. The subject suffers from any other eye disease(s) or other causes for the reduced visual acuity, aside from myopia and/or astigmatism.
2. The subject suffers from myopia-related visual complications resulting in visual loss, including myopic macular degeneration, myopic cataract and previous or pre-existing myopic retinal detachment.
3. The subject is suffering from Diabetes Mellitus.
4. The subject has previously undergone a refractive surgery procedure in either eye.
5. The subject is or may be pregnant.
6. The subject has an activity limitation due to medical disorders (including migraines, seizure disorders, etc.), medications, or emotional status that might potentially impair the subject's ability to perform the treatment.

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2004-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tan, FRCS, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

REFERENCES:
- [Background] Polat U, Sagi D. Lateral interactions between spatial channels: suppression and facilitation revealed by lateral masking experiments. Vision Res. 1993 May;33(7):993-9. doi: 10.1016/0042-6989(93)90081-7. PMID 8506641
- [Background] Sagi D, Tanne D. Perceptual learning: learning to see. Curr Opin Neurobiol. 1994 Apr;4(2):195-9. doi: 10.1016/0959-4388(94)90072-8. PMID 8038576
- [Background] Polat U, Norcia AM. Neurophysiological evidence for contrast dependent long-range facilitation and suppression in the human visual cortex. Vision Res. 1996 Jul;36(14):2099-109. doi: 10.1016/0042-6989(95)00281-2. PMID 8776476
- [Background] Polat U, Mizobe K, Pettet MW, Kasamatsu T, Norcia AM. Collinear stimuli regulate visual responses depending on cell's contrast threshold. Nature. 1998 Feb 5;391(6667):580-4. doi: 10.1038/35372. PMID 9468134
- [Background] Lim KL, Fam HB. NeuroVision treatment for low myopia following LASIK regression. J Refract Surg. 2006 Apr;22(4):406-8. doi: 10.3928/1081-597X-20060401-20. PMID 16629076
- [Background] Polat U, Ma-Naim T, Belkin M, Sagi D. Improving vision in adult amblyopia by perceptual learning. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6692-7. doi: 10.1073/pnas.0401200101. Epub 2004 Apr 19. PMID 15096608
- See also: Singapore Eye Research Institute — http://www.seri.com.sg/
- See also: Neurovision Website — http://www.neuro-vision.com/